CLINICAL TRIAL: NCT00003675
Title: A Randomized Phase II Trial of Oral Topotecan Given Twice a Day for 5 Days or Once a Day for 10 Days to Patients With Myelodysplastic Syndromes (MDS)
Brief Title: Topotecan in Treating Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-19803; U10CA031946 (NIH); CLB-19803; CDR0000066776 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2004-07-22 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: refractory anemia; refractory anemia with ringed sideroblasts; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; de novo myelodysplastic syndromes; secondary myelodysplastic syndromes; refractory cytopenia with multilineage dysplasia; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Topotecan 5 days (Experimental): Patients receive intervention twice daily for 5 days
  Interventions: Drug: topotecan hydrochloride
- Oral Topotecan 10 days (Experimental): Patients receive intervention once daily for 10 days
  Interventions: Drug: topotecan hydrochloride

INTERVENTIONS:
Drug: topotecan hydrochloride — 1.2 mg/sq m twice a day for 5 days (Arm I) and once a day for 10 days (Arm II)

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Randomized phase II trial to study the effectiveness of topotecan in treating patients who have myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate complete or partial remission, hematologic improvement, and cytogenic response rate when oral topotecan is given twice a day for 5 days versus once a day for 10 days to patients with myelodysplastic syndromes. II. Evaluate the safety and toxicity of oral topotecan in these patients. III. Evaluate whether there are morphologic and/or cytogenetic subsets of the myelodysplastic syndromes that will respond optimally to this regimen. IV. Evaluate the change in the percentage of bone marrow blast cells in these patients during treatment. V. Evaluate the time to transformation to acute myeloid leukemia (AML) or death in this patient population.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to FAB subtype: 1. Refractory anemia with excess blasts 2. Refractory anemia with excess blasts in transformation 3. Chronic myelomonocytic leukemia 4. Refractory anemia, refractory anemia with ringed sideroblasts, and refractory cytopenia with multilineage dysplasia Patients are randomized to receive oral topotecan either twice daily for 5 days or once daily for 10 days. Courses are repeated every 21 days. Patients are evaluated for hematologic response after the initial 2 courses, and then every 4 courses. If a partial response or hematologic improvement is observed, treatment continues until disease progression to acute myeloid leukemia, relapse, death, or irreversible toxicity. Patients who achieve a complete response receive an additional 2 courses of therapy before discontinuation of protocol treatment. Patients are followed every 3 months for 2 years, then every year for an additional 3 years, and at time of progression.

PROJECTED ACCRUAL: A total of 90 patients (45 per arm) will be accrued for this study within 13 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Primary or therapy-related myelodysplastic syndrome: Refractory anemia with excess blasts Refractory anemia with excess blasts in transformation Chronic myelomonocytic leukemia Refractory anemia, refractory anemia with ringed sideroblasts, or refractory cytopenia with multilineage dysplasia These patients must also have one of the following criteria: Greater than 4 units of RBCs transfused within the past 3 months OR Platelet count less than 50,000/mm3 OR Neutrophil count less than 1,000/mm3 AND a recent infection requiring antibiotics

PATIENT CHARACTERISTICS: Age: Over 15 Performance status: 0-2 Life expectancy: Not specified Hematopoietic: See Disease Characteristics Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT no greater than 2 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL Other: Not pregnant or nursing Fertile patients must use effective contraception Free of any evidence of prior cancer for at least 12 months

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 1 month since prior interferon No prior hematopoietic growth factors or cytokines except epoetin alfa No concurrent epoetin alfa Chemotherapy: No prior topotecan No prior chemotherapy for this disease At least 12 months since prior chemotherapy for another disease No other concurrent chemotherapy Endocrine therapy: At least 1 month since prior corticosteroids No concurrent hormonal therapy for disease-related conditions Concurrent steroids for adrenal failure allowed No concurrent dexamethasone and other steroidal antiemetics Radiotherapy: No prior radiotherapy for this disease At least 12 months since prior radiotherapy for another disease Surgery: Not specified Other: No prior cytotoxic therapy (including low-dose antimetabolites) for this disease At least 1 month since prior retinoids

Ages: 15 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 1999-03; Primary Completion 2002-01 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Response | During treatment and up to progression post treatment
  Response in the peripheral blood is assessed during tx, q 3 mon for 2 yrs post tx, then annually for another 3 years, and then at progression Bone marrow response is assessed prior to cycle 3, then q 4 cycles for the 1st yr. then q 8 cycles for patients who continue beyond
Toxicity | during treatment until progression
  assessment during treatment, q 3 mon for 2 years post tx, then annually for another 3 yrs, then at progression

CONTACTS AND LOCATIONS:
Overall Officials: David L. Grinblatt, MD, Study Chair — Louis A. Weiss Memorial Hospital
Locations (48):
- United States (48):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - University of California San Diego Cancer Center, La Jolla, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Illinois at Chicago Health Sciences Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Result] Klein CE, Kastrissios H, Miller AA, Hollis D, Yu D, Rosner GL, Grinblatt DL, Larson RA, Ratain MJ. Pharmacokinetics, pharmacodynamics and adherence to oral topotecan in myelodysplastic syndromes: a Cancer and Leukemia Group B study. Cancer Chemother Pharmacol. 2006 Jan;57(2):199-206. doi: 10.1007/s00280-005-0023-6. Epub 2005 Sep 13. PMID 16158312
- [Result] Grinblatt DL, Yu D, Hars V, et al.: Relationships of response to oral topotecan (Topo) for myelodysplastic syndrome (MDS) with IPSS group and cytogenetics - CALGB study 19803. [Abstract] Blood 100 (11 Pt 1): A-3137, 2002.
- [Result] Grinblatt DL, Yu D, Klein C, et al.: Two schedules of oral topotecan for myelodysplastic syndrome (MDS)-CALGB study 19803. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-1209, 2001.